CLINICAL TRIAL: NCT06576973
Title: A Prospective, Single-arm, Single-center, Exploratory Study of the Safety and Efficacy of Adbelimumab Combined With Chemotherapy and Apatinib in Patients With Resectable Esophageal Squamous Cell Carcinoma
Brief Title: Adbelimumab Combined With Chemotherapy and Apatinib in Patients With Resectable Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0949
Record Dates: First submitted 2024-08-25; First posted 2024-08-29 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Squamous Cell Carcinoma; Neoadjuvant Treatment
Keywords: Adbelimumab; Chemotherapy; Apatinib; Esophageal Squamous Cell Carcinoma; Neoadjuvant Treatment
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Carboplatin; apatinib; Esophagectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adbelimumab, chemotherapy and apatinib (Experimental): Preoperative neoadjuvant therapy for 4 cycles. Radical surgery is performed 4-6 weeks after the last dose. Postoperative radiotherapy is determined according to the clinical situation and pathological stage of the patient. Adbelimumab can be aintained for a maximum of 1 year. During the study, patients were be followed until disease progression, withdrawal of informed consent, loss of follow-up, or death.
  Interventions: Drug: Adbelimumab, Albumin paclitaxel, Carboplatin, Apatinib; Procedure: Esophagectomy; Other: Collecting samples from participant

INTERVENTIONS:
Drug: Adbelimumab, Albumin paclitaxel, Carboplatin, Apatinib — Adbelimumab 1200mg Day 1; Albumin paclitaxel 260mg/m2, Day 1; carboplatin AUC=5, Day 1; Apatinib 250mg Po Day 2-4. Preoperative neoadjuvant therapy for 4 cycles, one cycle every 21 days.
  Other Names: Esophagectomy
Procedure: Esophagectomy — Prior to each surgical procedure, the department engaged in comprehensive discussions and deliberations to ascertain and establish the most suitable course of action. Minimally invasive IvorLewis (intrathoracic anastomosis) or McKeown (neck anastomosis) esophagectomy, including two field extensive lymphadenectomies, was performed according to the tumor location. The resection length should be at least 5cm from the tumor origin according to prechemotherapy by endoscopy. The surgeries will be performed by surgeons with rich experience. Minimally invasive esophagectomy, can be performed using the da Vinci surgical robot, thoracoscope, or laparoscope, or by using an open approach, as judged appropriate by the surgeon.
Other: Collecting samples from participant — Blood, Tumour will be Collected from participant. Fate of sample is Destruction after use. 20 ml of peripheral blood was collected the day before each of the immunotherapy sessions and after surgery. Tumour sample will be collected before neoadjuvant therapy and after surgery.

SUMMARY:
Esophageal cancer is a prevalent digestive tract tumor, with around 400,000 new cases and 300,000 deaths globally each year. In the past few decades, surgery, radiotherapy, chemotherapy and other treatments were continuously improved, however, the mortality of esophageal squamous cell carcinoma (ESCC) patients was not significantly decreased. For patients with locally advanced esophageal cancer, direct surgery is not effective. It is difficult to achieve radical resection by surgery merely, and even if many patients receive surgery, they may eventually have tumor recurrence and poor survival rate.

Therefore, it is necessary to explore effective perioperative neoadjuvant treatment to reduce the risk of postoperative recurrence and improve the postoperative survival rate of patients. According to the reports, the expression of PD-L1 in esophageal cancer was about 41.4%. Therefore, PD-1/ PD-L1 immunocheckpoint inhibitor may become a new method for the treatment of ESCC. Preliminary clinical results showed that immunotherapy combined with chemoradiotherapy provided a synergies antitumor effect.

The results of the Phase 1b trial evaluating adbelimumab monotherapy as a neoadjuvant treatment for locally advanced resectable ESCC demonstrated that patients receiving two cycles of neoadjuvant sequential surgery exhibited favorable safety profiles, with no adverse reactions of grade 3 or higher. The trial reported a major pathological response (MPR) rate of 24%, a pathological complete response (pCR) rate of 8%, a 2-year overall survival (OS) rate of 92%, and a 2-year recurrence-free survival (RFS) rate of 100%. The effectiveness of combining adbelizumab with chemotherapy and targeted therapy for locally advanced esophageal cancer is uncertain.

This study aims to assess the efficacy and safety of using adbelizumab with chemotherapy and apatinib as neoadjuvant therapy for resectable ESCC.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Patients age 18 to 75 years old.
3. Primary resectable, histologically confirmed esophageal squamous cell cancer.
4. Esophageal squamous cell carcinoma the clinical stage was II-IVA (according to AJCC TNM stage, 8th edition).
5. ECOG PS 0-1.
6. No distant metastasis, the diseases could be resectable assessed by thoracic oncologist.

Exclusion Criteria:

1. With significant cardiovascular disease.
2. Current treatment with anti-viral therapy or HBV.
3. Female patients who are pregnant or lactating.
4. History of malignancy within 5 years prior to screening.
5. Active or history of autoimmune disease or immune deficiency.
6. Signs of distant metastases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (PCR) | 1 month after surgery
  The pCR will be defined as the proportion of participants with absence of residual tumor in the resected primary tumor and all resected lymph nodes after completion of neoadjuvant treatment.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | 1 month after surgery
  The MPR will be defined as the proportion of participants with less 10% of residual tumor in the resected primary tumor and all resected lymph nodes after completion of neoadjuvant treatment.
Objective Response Rate (ORR) | before surgery
  The ORR will be defined as the proportion of participants who have a complete response or partial response before surgery as assessed by the investigator per RECIST v1.1 in all participants with measurable disease at baseline
The changes in the peripheral blood immunoprofile and tumor tissue sample among non-PCR (NPCR) and PCR patients | 3 months after surgery
  By using mass spectrometry (CyTOF) and single-cell analysis, we comprehensively characterized the immune landscape in the peripheral blood and tumor sample of ESCC patients before and after anti-PD-1 immunotherapy, aiming to explore the immune subsets correlated with neoadjuvant immunotherapy response.
2-year and 5-year overall survival | 2-year and 5-year after enrolled
  The proportion of all study cases in which no death from any cause occurred within 2 years and 5 years after enrolled
Incidence of Treatment-related Adverse Events | 1 month after surgery
  Incidence of Treatment-related Adverse Events as Assessed by CTCAE v5.0
R0 resection rate | 1 month after surgery
  This will be defined as the proportion of participants with R0 resection

CONTACTS AND LOCATIONS:
Overall Officials: Wang, Study Chair — 2nd Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, China, China